CLINICAL TRIAL: NCT03807362
Title: A Single Center, Open Label Pilot Study to Evaluate the Safety and Efficacy of CC-11050 in Nepalese Patients With Erythema Nodosum Leprosum
Brief Title: CC-11050 Trial in Nepalese Patients With Erythema Nodosum Leprosum
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leprosy Mission Nepal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nepal CC-11050
Record Dates: First submitted 2018-09-14; First posted 2019-01-16 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Erythema Nodosum Leprosum; Leprosy
MeSH Terms: conditions — Leprosy | interventions — CC-11050

STUDY DESIGN:
Intervention Model Description: A single center, open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC-11050 treatment (Experimental): 200mg CC-11050 will be administered twice daily as a pill taken with food (at breakfast and evening meal) for participants with moderate to severe ENL for 10 days, then up to 28 days (during Step 1) and then up to 1 year (during Step 2).
  Interventions: Drug: CC-11050

INTERVENTIONS:
Drug: CC-11050 — CC-11050 is a novel anti-inflammatory compound with potential to treat a variety of chronic inflammatory conditions.

SUMMARY:
This study will be a single center, Phase 2, open-label trial to evaluate the safety and efficacy of 200mg CC-11050 administered twice daily taken with food for patients with moderate to severe ENL. The study will be performed in two steps: 1) to evaluate immediate effect in safety and efficacy of drug in 10 males with new or new recurrent episode ENL and, if found to be safe and effective by the DSMB and 2) if allowed by the DSMB, and approved by relevant study stakeholders, an additional 40 ENL patients will be enrolled for up to 52 weeks of treatment. A safety analysis will be conducted on all patients who have received at least one dose of study drug, and will include the frequency of all adverse events and laboratory abnormalities as well as frequency of dose interruptions, dose reductions and treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

Study participants must satisfy the following criteria to be enrolled in the study:

1. Must be 18 -65 years old, weight > 35kg for women and >40kg for men at the time of signing the informed consent.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Have signs or symptoms of new or new episode ENL. In Step one, participants must be male. In Step 2, participants can be either male or female.
4. Able to adhere to the study schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participants from participating in the study.
2. Patients on continuous rifampicin will be excluded, however, If rifampicin is given only once a month as part of a multi-drug regimen, a minimum of 2-week washout period is required prior to administration of CC-11050
3. Any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he were to participate in the study.
4. Any condition that confounds the ability to interpret data from the study (ie, HIV, chronic HepB, chronic HepC or TB patients under active treatment). Resolved TB patients will not be excluded from the study.
5. Stable and well managed patients with Diabetes and hypertension will not be excluded from the study.
6. Use of systemic corticosteroid or immunosuppressant therapy within 7 days of study medication initiation
7. Pregnant or nursing females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only for Step 1 (first 10 patients for testing up to 28 days of treatment). If successful, then both males and females can enroll in the second part of the study (up to 40 patients testing up to 1 year of therapy).
Enrollment: 50 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with moderate to severe ENL with severity changes as assessed by the ENL Severity Scale. | 10 days, 28 days and monthly up to 1 year of treatment
  Changes in ENL Severity Scale Score (Walker et al., PLoS Negl Trop Dis 11(7): e0005716, https://doi.org/10.1371/journal.pntd.0005716) as compared to baseline and any previous time points. Ten clinical categories contribute 0-3 points toward the total score of 0-30. An ENL patient with a total scale score of less than 9 is considered to have mild ENL, while scores >9 are considered moderate to severe ENL. A minimum score of 9 is required to indicate sufficient ENL symptoms from which post-intervention reduction in score(s) can be determined meaningful improvement.

SECONDARY OUTCOMES:
Number of participants with moderate to severe ENL with decreased duration of episode(s) as assessed by standard ENL episode definition. | 10 days, 28 days, monthly up to 1 year of treatment and up to 1 year followup after treatment cessation.
  Changes in ENL episode duration(s) as compared to baseline and any previous time points. By definition, if ENL symptoms are separated by time and no need of treatment for >28 days, they are considered separate episodes. Recurrence is anytime another episode occurs after >28 days of no prior treatment or symptoms.
Number of participants with moderate to severe ENL with decreased bacterial index (BI) as assessed by slit skin smear microscopy. | Enrolment and after 1 year treatment.
  Changes in slit skin smear microscopy BI as compared to baseline. BI can range from 0-6.
Number of participants with moderate to severe ENL with decreased bacterial index (BI) as assessed skin histopathology. | Enrolment and after 1 year treatment.
  Changes in skin histopathology bacterial index (BI) as compared to baseline. BI can range from 0-6.
Number of patients with moderate to severe ENL with improved peripheral neuropathy as assessed by standardized monofilament and voluntary muscle tests. | enrolment, 10 days, 28 days, biweekly (as needed), up to 1 year treatment, up to 1 year followup after treatment cessation
  Changes in scores for peripheral neuropathy as indicated by monofilament and voluntary muscle tests compared from baseline and any previous time points. To check neuropathy, 7 motor function nerves and 6 sensory function nerves on each side of the body are assessed for a total 26 nerves. Each are assessed on 3 sites using a standard set of Semmes-Weinstein monofilaments. The 200mg filament and the 2g filament represent threshold for the hand and foot, respectively. The 0-5 Medical Research Council (MRC) scale is used for motor function assessment. Sensory scores >3 and motor nerve scoring (MRC) < 5 are regarded impaired (indicating neuropathy). More method specifics can be found here: van Veen N.H., et al., Corticosteroids for treating nerve damage in leprosy. Cochrane Database Syst Rev, 2007(2): p. CD005491.
Number of participants with moderate to severe ENL with improved quality of life as assessed by the World Health Organization Quality of Life tool. | Enrolment, 28 days, monthly up to 1 year of treatment and up to 1 year followup after treatment cessation.
  Changes in scores for the World Health Organization Quality of Life assessment as compared to baseline and any previous time points. There are 26 questions in this questionnaire and each can be scored from 1 to 5 points. The highest possible score is 130 and lowest possible score is 26. A higher score denotes better quality of life.
Number of participants with moderate to severe ENL as assessed by standard blood panel and basic metabolic testing. | Enrolment, day 10, day 17, day 28, monthly up to 1 year of treatment, and 1 month post-cessation of treatment.
  Abnormalities or change in values in comparison to baseline and any previous time points.
Number of participants with moderate to severe ENL as assessed by urinalysis. | Enrolment, day 10, day 17, day 28, monthly up to 1 year of treatment, and 1 month post-cessation of treatment.
  Detection of albumin (qualitative) as compared to baseline and any previous time points. Urine albumin is related to ENL severity and kidney function test.
Number of participants with moderate to severe ENL as assessed by serological indicators associated with ENL. | Enrolment, day 10, day 17, day 28, monthly up to 1 year of treatment, and 1 month post-cessation of treatment.
  Detection of rheumatoid arthritis factor (positive) and/or C-reactive protein (positive) as compared to baseline and any previous time points.

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Shah, MD, Principal Investigator — The Leprosy Mission Nepal
Locations (2):
- Nepal (2):
  - The Leprosy Mission Nepal, Kathmandu, Bagmati
  - Anandaban Hospital, Lalitpur, Bagmati

IPD SHARING:
Plan to Share IPD: Undecided